CLINICAL TRIAL: NCT00194207
Title: Risk Factors as Predictors of Ectopic PRegnancy
Brief Title: Risk Factors of Ectopic Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Kurt T Barnhart, MD, MSCE, University of Pennsylvani
Other Study IDs: 103700; R01HD036455-01A1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify elements of a patient's demographics, history, and clinical presentation that may aid in differentiating between patients with an ectopic pregnancy, miscarriage, or normal intrauterine pregnancy. This study will also evaluate serial levels of human chorionic gonadotropin in the serum of these patients, as another way to make the diagnosis.

DETAILED DESCRIPTION:
The backbone of this protocol is the systematic evaluation of the presentation, work up, diagnosis and treatment outcome of women who present for evaluation of pain or bleeding in the first trimester of pregnancy and are therefore at risk for ectopic pregnancy (EP). Our focus is women whose diagnosis was not definitive upon initial presentation. We plan to collect systematic data regarding the current diagnostic strategies and treatment of these women and compare actual outcomes to those predicted by our newly developed strategies. This will be the first time such an endeavor has been conducted at multiple centers concomitantly. Expansion to two other sites is vital to ensure our preliminary data is valid and generalizable to women from different races and ethnicities, as well as to achieve the precision necessary to develop an accurate clinical tool. We will use a secure web-based clinical database (the Quantbook) to compile clinical information, and will download de-identified data to the research database once the diagnosis and clinical course of a patient has been completed. The Quantbook will be an expansion of a clinical database successfully utilized at Penn for the past 15 years. For a more detailed description of the Quantbook and research databases please see Attachment 2 of the full protocol. High quality information obtained from this cohort of women will allow the optimization and validation of our currently derived and proposed methods of diagnosis.

Data Collection Clinical Database (Quantbook): The clinician (e.g., attending physician, fellow, resident physician, nurse practitioner) who assesses the patient input information into the Quantbook. At the first presentation, this will include the patient's medical history, as well as presenting signs and symptoms. Results of tests ordered, including hCG and relevant chemistry, hematology, blood type, and ultrasound, will be entered. The clinician will assign a clinical impression (which may be a final definitive diagnosis, or a suspected diagnosis, or "unable to determine"). Follow-up contacts and assessments are recorded as they occur. Each time the patient returns for an assessment, the clinical impression can be updated, until a definitive diagnosis is made. A research coordinator will be tasked to monitor the Quantbook to provide quality control that the clinical data entered is complete and correct.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive-aged women
* Currently pregnant based on serum human chorionic gonadotropin test
* Present for care for vaginal bleeding and/or pelvic pain
* Final diagnosis of:

  1. Ectopic pregnancy
  2. Miscarriage less than 14 weeks gestation
  3. Ongoing normal intrauterine pregnancy less than 14 weeks gestation
* Entered into clinical tracking database

Exclusion Criteria:

* Patients not entered in clinical tracking database, or with insufficient information recorded to analyze (e.g. missing final diagnosis)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with early pregnancy with symptoms of pain and bleeding, presenting to the ER at the Hospital of University of Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 1999-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States